CLINICAL TRIAL: NCT02230657
Title: A Prospective, Randomized Trial Comparing Same Day Discharge and Overnight Hospital Stay Among Total Hip Arthroplasties Done by the Direct Anterior Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Collaborators: The Anderson Orthopaedic Clinic (Unknown)
Responsible Party: Sponsor
Other Study IDs: WHOZ01
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Osteoarthritis of the Hip
MeSH Terms: conditions — Osteoarthritis, Hip

ARMS (2):
- Same day Discharge (Active Comparator)
  Interventions: Procedure: Same day discharge
- Next day discharge (Active Comparator)
  Interventions: Procedure: Next day discharge

INTERVENTIONS:
Procedure: Same day discharge
  Arms: Same day Discharge
Procedure: Next day discharge
  Arms: Next day discharge

SUMMARY:
The purpose of this study is to identify differences in satisfaction, pain and length of stay between patients undergoing hip replacement who are discharged from the hospital on the day of surgery compared to patients who stay one night in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Primary THA without acute hip fracture or prior hardware that would need to be removed at the time of surgery
* Unilateral THA
* Pre-operative Body Mass Index (BMI) < 40 kg/m2
* Age < 75 years at time of surgery
* Pre-operative hemoglobin > 10 g/dL if pre-operative hemoglobin data is available
* No history of cardiopulmonary disease that would necessitate inpatient monitoring after surgery
* Pre-operative ambulatory status does not require the use of a walker or wheelchair
* No chronic pre-operative opioid medication use or opioid addiction
* Assistance available at home after discharge from hospital
* No other condition or circumstance that would preclude rapid discharge from the hospital after surgery
* Subject's English proficiency allows understanding of study and Informed Consent
* Subject consented to participate in this study

Exclusion Criteria:

* Revision THA
* Bilateral THA
* Pre-operative BMI ≥ 40 kg/m2
* Age ≥ 75 at time of surgery
* Pre-operative hemoglobin ≤ 10 g/dL if pre-operative hemoglobin data is available
* History of cardiopulmonary disease requiring acute inpatient monitoring
* Pre-operative ambulatory status requiring the use of a walker or wheelchair
* Chronic pre-operative opioid medication use or opioid addiction
* Limited or no assistance available at home after discharge from hospital
* Any other condition or circumstance that would preclude rapid discharge from the hospital
* Subject not proficient in English
* Subject did not consent to participate in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | Discharge through 30 days post-op

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rothman Institute, Philadelphia, Pennsylvania
  - The Anderson Orthopaedic Clinic, Alexandria, Virginia